CLINICAL TRIAL: NCT06360926
Title: Improvement Image Quality for SuperSonic® MACH Ultrasound System
Acronym: MACH IQ
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of the study
Sponsor: SuperSonic Imagine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A00526-41
Record Dates: First submitted 2024-03-19; First posted 2024-04-11 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- SuperSonic® Ultrasound System equipped with new software iterations used with a new probe (Experimental)
  Interventions: Device: SuperSonic® Ultrasound System

INTERVENTIONS:
Device: SuperSonic® Ultrasound System — SuperSonic® Ultrasound System equipped with new software iterations used with a new probe and CE marked probes. The new software and probe are the new study investigational device not CE marked

SUMMARY:
The aim of this Study is to collect radiologist feedback to support the further development and improvement of the imaging modes implemented on the embedded software in the SuperSonic® Ultrasound System (including the probe).

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years old and is able to understand and sign the informed consent form.
* Subject is a minor < 18 years old and the legal representative has signed the informed consent form.
* Subject is scheduled for at least one or more routine ultrasounds.
* Subject is affiliated to National Social Insurance or a Health Insurance Regimen.

Exclusion Criteria:

* Subject is unable or unwilling to adhere to Study procedures.
* Subject or his/her legal representative if a minor is unable to express or understand informed consent.
* Subject is under legal protection
* Subject is deprived of liberty by judicial or administrative decision
* Subject undergoes psychiatric treatment under constraint
* Subject is admitted to a health or social establishment for purposes other than research
* Subject has latex allergy.
* Subject has an open wound, cut, and/or a rash which would preclude an ultrasound imaging procedure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of image quality | During ultrasound procedure
  Following the two ultrasound procedures, the radiologist will rate the image quality produced by the Study Device, compared to that produced by the SOC ultrasound. A score from 1 to 5 (1: Not acceptable; 2: Acceptable; 3: Fair; 4: Good; 5: Excellent) for each of the characteristics of the image: General Aesthetics; Spatial Resolution; Contrast Resolution; Temporal Resolution; Penetration and Sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Necker-Enfants malades, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No